CLINICAL TRIAL: NCT03508570
Title: Phase Ib Clinical Investigation of Intraperitoneal Ipilimumab and Nivolumab in Patients With Peritoneal Carcinomatosis Due to Gynecologic Cancers
Brief Title: Nivolumab With or Without Ipilimumab in Treating Patients With Recurrent or High Grade Gynecologic Cancer With Metastatic Peritoneal Carcinomatosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017-0264; NCI-2018-00282 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2017-0264 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2018-04-16; First posted 2018-04-25 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Malignant Peritoneal Neoplasm; Malignant Retroperitoneal Neoplasm; Metastatic Cervical Carcinoma; Metastatic Endometrial Carcinoma; Metastatic Fallopian Tube Carcinoma; Metastatic Malignant Female Reproductive System Neoplasm; Metastatic Ovarian Carcinoma; Metastatic Primary Peritoneal Carcinoma; Peritoneal Carcinomatosis; Platinum-Refractory Fallopian Tube Carcinoma; Platinum-Refractory Malignant Female Reproductive System Neoplasm; Platinum-Refractory Ovarian Carcinoma; Platinum-Refractory Primary Peritoneal Carcinoma; Platinum-Resistant Fallopian Tube Carcinoma; Platinum-Resistant Malignant Female Reproductive System Neoplasm; Platinum-Resistant Ovarian Carcinoma; Platinum-Resistant Primary Peritoneal Carcinoma; Recurrent Cervical Carcinoma; Recurrent Endometrial Carcinoma; Recurrent Fallopian Tube Carcinoma; Recurrent Malignant Female Reproductive System Neoplasm; Recurrent Ovarian Carcinoma; Recurrent Primary Peritoneal Carcinoma; Stage IV Fallopian Tube Cancer AJCC v8; Stage IV Ovarian Cancer AJCC v8; Stage IV Primary Peritoneal Cancer AJCC v8; Stage IVA Fallopian Tube Cancer AJCC v8; Stage IVA Ovarian Cancer AJCC v8; Stage IVA Primary Peritoneal Cancer AJCC v8; Stage IVB Cervical Cancer AJCC v8; Stage IVB Fallopian Tube Cancer AJCC v8; Stage IVB Ovarian Cancer AJCC v8; Stage IVB Primary Peritoneal Cancer AJCC v8; Stage IVB Uterine Corpus Cancer AJCC v8
MeSH Terms: conditions — Uterine Cervical Neoplasms; Endometrial Neoplasms; Fallopian Tube Neoplasms; Ovarian Neoplasms; Peritoneal Neoplasms | interventions — Ipilimumab; CTLA-4 Antigen; Nivolumab; Pharmacogenomic Variants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group I (nivolumab) (Experimental): Patients receive nivolumab i.p. over 90 minutes on days 1, 15, and 29. Cycles repeat every 6 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Biological: Nivolumab; Other: Pharmacokinetic Study
- Group II (nivolumab and ipilimumab) (Experimental): Patients receive nivolumab as in group I and ipilimumab i.p. on day 1. Cycles repeat every 6 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Ipilimumab; Other: Laboratory Biomarker Analysis; Biological: Nivolumab; Other: Pharmacokinetic Study

INTERVENTIONS:
Biological: Ipilimumab — Given i.p.
  Other Names: Anti-Cytotoxic T-Lymphocyte-Associated Antigen-4 Monoclonal Antibody; BMS-734016; Ipilimumab Biosimilar CS1002; MDX-010; MDX-CTLA4; Yervoy
  Arms: Group II (nivolumab and ipilimumab)
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Nivolumab — Given i.p.
  Other Names: BMS-936558; CMAB819; MDX-1106; NIVO; Nivolumab Biosimilar CMAB819; ONO-4538; Opdivo
Other: Pharmacokinetic Study — Correlative studies
  Other Names: PHARMACOKINETIC; PK Study

SUMMARY:
This phase Ib trial studies the side effects and best dose of nivolumab with or without ipilimumab in treating patients with female reproductive cancer that has come back (recurrent) or is high grade and has spread extensively throughout the peritoneal cavity (metastatic). Immunotherapy with monoclonal antibodies, such as nivolumab and ipilimumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the recommended phase II dose (RP2D) of intraperitoneal (i.p.) nivolumab in combination with ipilimumab.

SECONDARY OBJECTIVES:

I. To describe the pharmacokinetics (PK), toxicities, and immune-related adverse events associated with i.p. checkpoint inhibitor therapy.

II. To estimate the clinical benefit rate (rate of partial response [PR], complete response [CR], and stable disease [SD] using Response Evaluation Criteria in Solid Tumors [RECIST] version 1.1 modified to include immune-related response criteria) for the expansion cohort.

EXPLORATORY OBJECTIVES:

I. To determine blood based transcriptional changes associated with pharmacokinetics (PK) time points and determine their correlation with serum drug concentrations, clinical response, and immune related adverse events.

II. To determine baseline and on-treatment molecular alteration (ribonucleic acid [RNA] and protein) associated with i.p. and nivolumab (Nivo) (for the expansion cohort).

OUTLINE: This is a dose-escalation study. Patients are assigned to 1 of 2 groups.

GROUP I: Patients receive nivolumab i.p. over 90 minutes on days 1, 15, and 29. Cycles repeat every 6 weeks in the absence of disease progression or unacceptable toxicity.

GROUP II: Patients receive nivolumab as in group I and ipilimumab i.p. on day 1. Cycles repeat every 6 weeks in the absence of disease progression or unacceptable toxicity.

After completion of the study treatment, patients are followed up every 6 weeks for at least 100 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have biopsy-confirmed ovarian or other gynecologic cancers (fallopian tube, peritoneal, endometrial, or cervical cancer) who have recurred after or progressed on frontline and one or more second-line standard treatments; patients with ovarian/fallopian tube/peritoneal cancers must have platinum refractory or resistant disease (defined as progression on a platinum containing regimen or recurrence within 180 days of prior dose of platinum-containing regimen), but do not require second-line treatment to be eligible for the dose-finding phase; eligibility for the expansion cohort will be limited to subjects with high grade epithelial ovarian, fallopian tube, or peritoneal carcinomas who have recurred after or progressed on frontline and one or more second-line standard treatments or have developed platinum resistant disease after frontline therapy (in which case progression on a second line therapy will not be required); however, for the dose expansion phase, potential subjects are not required to have platinum refractory or resistant disease
* Measurable metastatic disease (by RECIST version [v] 1.1) in the peritoneal cavity or retroperitoneal lymph nodes; disease outside of the peritoneal cavity is allowed as long as metastatic sites are also present within the peritoneum/retroperitoneum
* Absolute neutrophil count >= 1500/mL
* Platelets >= 100,000/mL
* Hemoglobin >= 9 g/dL (transfusion to meet this criterion is allowed)
* Serum creatinine clearance (CL) >= 40 mL/min by the Cockcroft-Gault formula (Cockcroft and Gault 1976) or by 24-hour urine collection for determination of creatinine clearance
* Total bilirubin =< 1.5 X upper limit of normal (ULN)
* Aspartate aminotransferase (AST/serum glutamic-oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT/serum glutamate pyruvate transaminase [SGPT]) =< 2.5 X ULN (=< 5 X ULN in subjects with bone or liver metastases)
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 or 1
* Subjects must be >= 4 weeks beyond treatment with any chemotherapy or other investigational therapy to include hormonal, biological, or targeted agents (>= 8 weeks from previous bevacizumab treatment) at the time of first dose of study drug(s)
* Women of child-bearing potential MUST have a negative serum human chorionic gonadotropin (HCG) test unless prior hysterectomy or menopause (defined as 12 consecutive months of amenorrhea); subjects are considered not to be of child-bearing potential if they are surgically sterilized or post-menopausal (>= 50 years of age and has not had menses for greater than 1 year or with serum follicle stimulating hormone [FSH] in the menopausal range will be considered postmenopausal); subjects should not become pregnant or breastfeed while on this study; sexually active subjects of child bearing potential must agree to use contraception for the duration of study participation and for 5 months after the last dose of ipilimumab or nivolumab
* Ability to understand and willingness to sign informed consent form prior to initiation of the study and any study procedures
* Subjects in expansion cohort only: Willing to undergo pre- and on-treatment biopsies

Exclusion Criteria:

* Patients who are pregnant or breastfeeding
* Patients with low grade ovarian/fallopian tube/peritoneal cancers
* Prior immune checkpoint inhibitor therapy
* History of inflammatory bowel disease (including ulcerative colitis and Crohn's disease), or any other known autoimmune diseases including rheumatoid arthritis, scleroderma, systemic lupus erythematosus, and autoimmune vasculitis
* History of previous malignancy that in the principal investigator (PI)'s opinion has a reasonable chance of recurrence during the study period or otherwise confounding this clinical trial
* Active peritonitis or diverticulitis
* Patients requiring corticosteroids use at doses greater than prednisone 10 mg daily equivalent (use of inhaled steroids, and short-term steroid for radiologic contrast allergy, or treatment of immune-related adverse events are allowed)
* Medical or surgical history that in the treating physician's opinion would make the subject not a suitable candidate for i.p. therapy; examples would include surgically documented extensive intraperitoneal adhesions or large volume ascites
* History of chronic obstructive pulmonary disease (COPD) or other chronic pulmonary disease requiring systemic steroid therapy, oxygen, or hospitalization
* Chronic hepatitis B or C virus infection, or known human immunodeficiency virus (HIV) positive, that might affect host immunity
* Any other illness or condition that in the investigator's opinion would adversely affect the safety of checkpoint inhibitor therapy
* Active infection requiring intravenous (IV) antibiotics or other uncontrolled intercurrent illness requiring hospitalization
* Inability to comply with the study and follow-up procedures
* History of cerebrovascular accident, myocardial infarction or unstable angina within the previous 6 months before starting therapy
* Prolongation of QT interval (QT)/corrected QT interval (QTc) (QTc interval > 470 ms) using the Fridericia method of QTc analysis
* Known active central nervous system metastases and/or carcinomatous meningitis
* History of severe hypersensitivity reaction with biologics therapy (monoclonal antibodies)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2018-09-21 (Actual); Primary Completion 2024-11-11 (Actual); Study Completion 2024-11-11 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD)/recommended phase II dose (RP2D) of intraperitoneal (i.p.) nivolumab in combination with ipilimumab | 12 weeks
  The RP2D or the MTD is defined as the combination of ipilimumab + nivolumab with the dose limiting toxicity (DLT) rate =< 30%. Dose-finding for the combination of ipilimumab plus nivolumab will be done using the data-augmentation continuous reassessment method (DA-CRM).

CONTACTS AND LOCATIONS:
Overall Officials: Amir A Jazaeri, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Background] Knisely A, Hinchcliff E, Fellman B, Mosley A, Lito K, Hull S, Westin SN, Sood AK, Schmeler KM, Taylor JS, Huang SY, Sheth RA, Lu KH, Jazaeri AA. Phase 1b study of intraperitoneal ipilimumab and nivolumab in patients with recurrent gynecologic malignancies with peritoneal carcinomatosis. Med. 2024 Apr 12;5(4):311-320.e3. doi: 10.1016/j.medj.2024.02.003. Epub 2024 Mar 11. PMID 38471508
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org